CLINICAL TRIAL: NCT03390803
Title: Effect of Hemifacial Spasm on Intraocular Pressure Measurement
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Funda Dikkaya, Medical Doctor, Medipol University
Other Study IDs: 02-115621
Record Dates: First submitted 2017-12-26; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Hemifacial Spasm; Intraocular Pressure
MeSH Terms: conditions — Hemifacial Spasm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with hemifacial spasm
  Interventions: Other: effect of hemifacial spasm on intraocular pressure
- healthy control subjects
  Interventions: Other: effect of hemifacial spasm on intraocular pressure

INTERVENTIONS:
Other: effect of hemifacial spasm on intraocular pressure — To evaluate the effect of Hemifacial spasm on Intraocular pressure measurement.

SUMMARY:
Twenty-four consecutive patients with Hemifacial spasm and 25 age and gender-matched randomly selected eyes of healthy volunteers underwent corneal pachymetry and intraocular pressure measurements using Goldmann Applanation Tonometer and non-contact tonometer. An interval of 15 minutes was maintained between Goldmann Applanation Tonometer and non-contact tonometer measurements. Intraocular pressure measurements were performed before (during hemifacial spasm) and 2 weeks after Botox injections in Hemifacial spasm patients and in healthy volunteers without Botox injections. All the measurements with Goldmann Applanation Tonometer were carried out by a single physician while those with the non-contact tonometer were done by another physician who was masked to the results of the Goldmann Applanation Tonometer. All measurements were taken between 10:00 and 11:00 a.m.

ELIGIBILITY:
Inclusion Criteria:

* patients with hemifacial spasm

Exclusion Criteria:

* Subjects will be excluded if they have allergies to botulinum toxin or any component of the drug, previous eyelid, refractive or intraocular surgery, any abnormality preventing reliable tonometry in either eye, strabismus, contact lens wear, pregnancy, glaucoma, ocular hypertension and patients using agents that could interfere with neuromuscular transmission.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty-four consecutive patients with Hemifacial spasm (study group) and twenty-five age-matched and gender-matched healthy volunteers (control group) will be prospectively included in the study. Intraocular pressure measurements will be performed before and 2 weeks after Botox injections in patients with HFS (involved and uninvolved eyes of HFS both) and in healthy volunteers without Botox injections.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Effect of Hemifacial Spasm on Intraocular Pressure Measurement Change | 2 week
  intraocular pressure measurements will be performed before and 2 weeks after Botox injections in patients with Hemifacial spasm (involved and uninvolved eyes of Hemifacial spasm both) and in healthy volunteers without Botox injections. The change between measurements will be evaluated.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cicik E, Yildirim R, Arici C, Dikkaya F, Arslan OS. Effect of Hemifacial Spasm on Intraocular Pressure Measurement. J Ophthalmol. 2018 Feb 6;2018:3621215. doi: 10.1155/2018/3621215. eCollection 2018. PMID 29545951